CLINICAL TRIAL: NCT00231075
Title: National, Phase II Study Designed to Evaluate the Safety and Efficacy of Paraplatin in Combination With Taxol in Patients of 70 Years and Older With Ovary Cancer F.I.G.O. Stages III and IV. FAG-2
Brief Title: Evaluation of the Safety and Efficacy of Paraplatin in Combination With Taxol in Patients of 70 Years and Older With Ovary Cancer F.I.G.O. Stages III-IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAG-2
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2005-11-03 (Estimated); Status verified 2005-09

CONDITIONS: Ovarian Cancer
Keywords: Epithelial ovary cancer F.I.G.O. stages III or IV; 70 years or older
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: Paraplatin
Drug: Paclitaxel

SUMMARY:
Safety and Efficacy of Paraplatin in combination with Taxol in patients of 70 years or older with epithelial ovary cancer F.I.G.O. stages III and IV.

DETAILED DESCRIPTION:
The Main objective of this study is to evaluate the faisibility of chemotherapy with Paraplatin in combination with Taxol in patients of 70 years or older with epithelial ovary cancer F.I.G.O. stages III and IV and to determine principal predictive factors of this feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven diagnosis of epithelial ovary cancer F.I.G.O stages III or IV (when only cytological proven diagnosis is available: malignant cells and pelvis tumoral mass and increased CA-125 must be diagnosed simultaneously)
* Patient aged > 70 years
* Neutrophil polynuclears > 1500/mm3 and Platelets > 100 000/mm3
* No clinical icterus
* Life expectancy of at least 3 months

Exclusion Criteria:

* Previous diagnosis of malignancy
* Previous chemotherapy treatment
* Previous radiotherapy
* Hypersensitivity to products containing Cremophore EL
* Hepatic values: bilirubine > 2*LSN, SGOT-SGPT > 2*LSN and/or Alkalin phosphatase > 3*LSN
* Myocardiopathy with arrhythmia

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75
Dates: Start 2001-01; Study Completion 2007-05

PRIMARY OUTCOMES:
Feasibility of the combination Paraplatine + Taxol (at least 6 cures have been administered for a given patient and for the treated population, 50% feasibility)

SECONDARY OUTCOMES:
Toxicity assessment
Overall survival
Progression-free survival
Rate of response
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Freyer, MD, PhD, Principal Investigator — Centre Hospitalier Lyon-Sud 69495 Pierre-Bénite cedex
Locations (2):
- France (2):
  - Centre Hosptalier Emile Roux, Eaubonne
  - Centre Hospitalier Lyon-sud, Pierre-Bénite